CLINICAL TRIAL: NCT04932876
Title: Assessment of the Response of the Immune System of Patients With End Stage Kidney Disease on Dialysis and Kidney Transplant Recipients Vaccinated for COVID-19
Brief Title: The Response of the Immune System of Patients With End Stage Kidney Disease on Dialysis and Kidney Transplant Recipients Vaccinated for COVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Ioannina (Other)
Responsible Party: Principal Investigator, Evangelia Ntounousi, Assistant Professor Of Nephrology, University of Ioannina
Other Study IDs: RESCOMUOI82152
Record Dates: First submitted 2021-05-19; First posted 2021-06-21 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: End Stage Kidney Disease; Kidney Transplantion; Covid19; Vaccination
Keywords: End Stage Kidney Disease; Kindey Trasplantation; Immune System; Covid19 Vaccination
MeSH Terms: conditions — Kidney Failure, Chronic; COVID-19 | interventions — COVID-19 Vaccines

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ESKD - HD: End Stage Kidney Disease on Long Term Dialysis
  Interventions: Biological: SARS - COV 2 VACCINE
- KTR: Kidney Transplant Recipient
  Interventions: Biological: SARS - COV 2 VACCINE

INTERVENTIONS:
Biological: SARS - COV 2 VACCINE — Vaccination for SARS - COV 2

SUMMARY:
Observational study of patients with End Stage Kidney Disease on dialysis and Kidney Transplant Recipients, before and after vaccination for SARS-COV 2, after written consent, with the aim of laboratory efficacy of the vaccine and safety regarding the clinical outcome of patients and possible complications.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Covid 19 vaccination

Exclusion Criteria:

* previous covid infection
* recent infection
* chronic infection
* HBV, HCV, HIV
* Active malignancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: End Stage Kidney Disease and Kidney Transplant Recipients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-04-24 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Efficacy of the vaccine | 24 months
  Humoral immune response to the vaccine as evaluated by generation of SARS-CoV-2 IgG II antibodies at two time points (before the second dose of the BNT162b2 vaccine and two weeks following the second dose of the BNT162b2 vaccine). Secondly, lympocyte subsets will be measured by flow cytometry (Naive and memeory T cells - CD45RO+, CD45 RA+, CD4+RO+, CD4+CDRA+, CD4+, CD8+, CD19+, NKT cells) at the two respective time points so as to assess alterations induced by vaccination. Serologic response will be estimated by measurement of anti SARS-CoV-2-spike IgGII titer (AU/ml) in the serum (using the ARCHITECT IgG II Quant test (Abbott); titers >50 arbitrary units (AU)/ml are considered positive (detection range, 6.8-80,000 AU/ml); positive agreement, 99.4%; negative agreement, 99.6%).

SECONDARY OUTCOMES:
Complications caused by the vaccine | 24 months
  Potential side effects associated with the vaccine shall be recorded. Percentages of lymphocytes subsets (as depicted before) in peripheral blood will be measured by flow cytometry. We will compare changes from baseline in the percentages of the lymphocytes subsets following the first and second dose of vaccination between the hemodialysis and kidney transplant recipeints group. In addition we will search for associations between percentages of lymphocytes subsets at diggerent measurement time points and antibody reponse.

CONTACTS AND LOCATIONS:
Locations (1):
- Evangelia Ntounousi, Ioannina, Epirus, Greece